CLINICAL TRIAL: NCT04660175
Title: The Efficacy and Safety of Non-resistance Manual Therapy in Inpatients With Acute Neck Pain Caused by Traffic Accidents: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2020-13
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Whiplash Injury of Cervical Spine
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-resistance therapy (Experimental): From the 2nd to 5th day of hospitalization, once a day, 4 times of non-resistance therapy is administered. And non-resistance therapy group is also treated with other Korean integrative medicine treatment everyday: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Other: non-resistance therapy; Other: acupuncture; Other: chuna; Other: pharmacoacupuncture; Drug: Korean herbal medicine
- Oriental medicine integrated treatment (Active Comparator): The control group is received Korean integrative medicine treatment everyday; acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Other: acupuncture; Other: chuna; Other: pharmacoacupuncture; Drug: Korean herbal medicine

INTERVENTIONS:
Other: non-resistance therapy — The non-resistance technique, created in Jaseng Hospital, is a combination of ischemic compression and mobilization It is a treatment that improves the limited range of motion of the cervical spine and relieves pain by applying ischemic pressure to the induration of the neck and at the same time firmly supporting the patient's head to give passive joint movements and completely relax.
  Arms: Non-resistance therapy
Other: acupuncture — According to the judgment of the oriental medicine doctor, select acupuncture point and tender spots such as BL10, TE14, GB20, GV16, etc. to a depth of 10 mm 6 -Self needle in 12 blood spots.
Other: chuna — Chuna treatment is administered once a day during the hospitalization period. Chuna is Korean manual therapy using methods such as joint mobilization, joint distraction, fascia relaxation and manipulation.
Other: pharmacoacupuncture — This is an oriental medical practice in which a certain amount of a drug extracted from a specific herbal medicine is injected with an injector to treat the patient's constitution, disease state, etc., and then injected into the treatment acupuncture points and body surface reaction points. Depending on the condition of the inpatient, acupuncture is used in parallel.
Drug: Korean herbal medicine — Formulated with herbal medicinal and pack the extract in a pouch, and have the hospitalized patient take it once in the morning and afternoon for 30 minutes after meals.

SUMMARY:
Non-resistance therapy is a combination of muscle compression relaxation technique and joint mobilization in patients with acute neck pain caused by traffic accidents. This study is to evaluate the effectiveness and safety of non-resistance therapy for pain and function problems in patients complaining of acute neck pain induced by traffic accidents.

So, investigators conduct a randomized controlled trials to verify the effectiveness and safety of non-resistance therapy. From December 2020 to May 2021, investigators recruit 120 inpatients who are suffered from acute neck pain with the numeric rating scale(NRS) over 5 by traffic accident(TA).

The Korean medical treatment group(n=60) receives daily acupuncture, herbal medicine, and chuna treatment as inpatient treatment from hospitalization until discharge. For the non-resistance therapy group(n=60), the korean medical treatment is performed in the same manner, but additional non-resistance therapy is performed once a day from the 2nd day to the 5th day of hospitalization.

Baseline is the time point before treatment for non-resistance therapy on the second day of hospitalization, and the primary endpoint is the time point after treatment on the 5th day (v5) after hospitalization.

For these two groups, investigators compare NRS(Numeric Rating Scale), Visual Analogue Scale(VAS), Range Of Motion(ROM), Neck Disability Index(NDI), the 12-Item Short Form Health Survey(SF-12), and PTSD Checklist for DSM(Diagnostic and Statistical Manual of Mental Disorders, DSM)-5(PCL-5).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-70 years on the date they sign the consent form
* Patients with NRS ≥ 5 for neck pain
* Patients who needs hospitalization due to acute neck pain that occurred within 7 days after traffic accident
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients with a specific serious disease that may cause acute neck pain: malignancy, fracture of lumbar spine, etc.
* Patients with progressive neurological deficits or with severe neurological symptoms
* The cause of pain is due to soft tissue disease, not the spine: tumors, fibromyalgia, rheumatoid arthritis, gout, etc.
* Patients with other chronic conditions that may interfere with the interpretation of the therapeutic effects or results: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study
* Patients who are pregnant, planning to become pregnant, or are breastfeeding
* Patients who have had surgery or procedures of cervical spine within the last three weeks
* Patients with a serious mental illness
* Patients who has not passed one month since the end of participation in other clinical studies, or plan to participate in other clinical studies during the study participation and follow-up period within 12 weeks
* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of neck pain | Change from baseline NRS at 5 days
  The extent of acute neck pain and discomfort was assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participants are asked to report their neck pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Numeric Rating Scale(NRS) of neck pain | baseline(day2), day3, day4, day5, day of Discharge(up to 14days), week 12
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participants are asked to report their neck pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'
Visual Analogue Scale (VAS) of neck pain | baseline(day2), day3, day4, day5, day of Discharge(up to 14days
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Visual Analogue Scale (VAS) of arm pain | baseline(day2), day3, day4, day5, day of Discharge(up to 14days)
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Numeric Rating Scale(NRS) of arm pain | baseline(day2), day3, day4, day5, day of Discharge(up to 14days), week 12
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10.
Range of movement (ROM) of flexion | baseline(day2), day3, day4, day5, day of Discharge(up to 14days)
  Range of movement (ROM) of flexion is measured.
Range of movement (ROM) of extension | baseline(day2), day3, day4, day5, day of Discharge(up to 14days)
  Range of movement (ROM) of extension is measured.
Range of movement (ROM) of left lateral flexion | baseline(day2), day3, day4, day5, day of Discharge(up to 14days)
  Range of movement (ROM) of left lateral flexion is measured.
Range of movement (ROM) of right lateral flexion | baseline(day2), day3, day4, day5, day of Discharge(up to 14days)
  Range of movement (ROM) of right lateral flexion is measured.
Range of movement (ROM) of left rotation | baseline(day2), day3, day4, day5, day of Discharge(up to 14days)
  Range of movement (ROM) of left rotation is measured.
Range of movement (ROM) of right rotation | baseline(day2), day3, day4, day5, day of Discharge(up to 14days)
  Range of movement (ROM) of right rotation is measured.
Neck Disability Index (NDI) | baseline(day2), day5, day of Discharge(up to 14days), week 12
  Functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range: 0 (better outcome) to 100 (worse outcome)
Patient Global Impression of Change (PGIC) | day5, day of Discharge(up to 14days), week 12
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.
12-item Short-Form Health Survey (SF-12) | baseline(day 2), day5, day of Discharge(up to 14days), week 12
  The SF-12 is a shortened version of the Short Form-36 Health Survey (SF-36), which is a widely used instrument to assess health-related quality of life. The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
Credibility and Expectancy | baseline(day 2)
  Credibility and Expectancy is a 9-point scale-likert-scale to evaluate the participants' expectations for treatment.(1 = not at all, 5 = somewhat, and 9 = very much)
Korean version of The Posttraumatic Stress Disorder Checklist for DSM-5(PCL-5-K) | baseline(day 2), day5, day of Discharge(up to 14days), week 12
  The PCL-5(The Posttraumatic Stress Disorder Checklist for DSM-5) is a 20-item, 5-point-Likert-scale, self-report questionnaire to measure the PTSD symptoms in the DSM-536 and to diagnose PTSD. A higher score (out of 80) indicates severe PTSD.
Drug Consumption | baseline(day2), day3, day4, day5, day of Discharge(up to 14days), week 12
  During the study period, the type and dose of drugs (prescribed due to the current medical history or remedy) were observed through a questionnaire when visiting the study subjects.
Adverse events | baseline(day2), day3, day4, day5, day of Discharge(up to 14days), week 12
  Safety outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Daejeon Jaseng Hospital of Korean Medicine, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi SW, Kim KH, Yoon JY, Lee SW, Park JW, Hong HW, Kyeong DH, Kim MK, Kim SN, Kim CY, Lee YJ, Lee JH, Kim JY, Ha IH. Effectiveness and safety of manual therapy for inpatients with traffic accident-induced acute neck pain: A randomized controlled trial. J Integr Med. 2026 Jan;24(1):81-89. doi: 10.1016/j.joim.2025.10.008. Epub 2025 Nov 1. PMID 41298158
- [Derived] Kim S, Kyeong DH, Kim MK, Kim CY, Lee YJ, Lee J, Ha IH, Park KS. The efficacy and safety of non-resistance manual therapy in inpatients with acute neck pain caused by traffic accidents: A randomized controlled trial. Medicine (Baltimore). 2022 Jun 3;101(22):e29151. doi: 10.1097/MD.0000000000029151. PMID 35665724